CLINICAL TRIAL: NCT02283944
Title: TMS Electrochemotherapy for Glioblastoma Multiforme
Status: Withdrawn | Phase: Phase 2 | Type: Interventional
Why Stopped: Device for multi coil TMS no longer supported
Sponsor: University of Aarhus (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 15102014
Record Dates: First submitted 2014-11-03; First posted 2014-11-05 (Estimated); Last update posted 2021-09-20 (Actual); Status verified 2014-10

CONDITIONS: Glioblastoma
MeSH Terms: conditions — Glioblastoma | interventions — Transcranial Magnetic Stimulation

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (1):
- TMS electrochemotherapy (Experimental): Combined TMS (transcranial magnetic stimulation) and Temozolomide chemotherapy.
  Interventions: Device: TMS

INTERVENTIONS:
Device: TMS — Pulsed non-invasive brain stimulation using electromagnets
  Other Names: Transcranial Magnetic Stimulation

SUMMARY:
The proposed project aims to develop novel electrochemotherapeutic treatment of glioblastoma multiforme (GBM). Standard treatment has limited effect on survival and quality of life. Electrochemotherapy is a novel and promising treatment, which has demonstrated convincing results in the treatment of various types of carcinoma. The treatment is based on a combination of electrical current stimulation of tumor cells and simultaneous administration of chemotherapeutic drugs. Electrochemotherapy works by inducing an electrical current between implanted electrodes in the tumor tissue, causing electroporation of the cancer cell membranes, and thereby increasing the cellular permeability and drug uptake. Electrochemotherapy has proven to be an efficient way of considerably increasing the potency of the chemotherapeutic drug bleomycin in malignant cells in skin tumors and carcinoma metastases, and thereby increasing cytotoxicity of the drug locally in the tumor tissue. This allows for treatment with lower doses of chemotherapeutic drugs and more defined, local area of effect, thus decreasing systemic effects. The investigators propose to use a novel non-invasive and safe technique called focused transcranial magnetic stimulation (focused TMS) to induce electrical current in the tumor tissue. TMS is a safe and widely implemented technology used to treat multiple neurological diseases such as pain, depression and stroke. Studies have shown that effective electroporation of cell membranes can be obtained using induction of electromagnetic fields in a cell suspension, and new focused TMS further enables focused treatment of selected brain regions without surgical intervention and, thereby focusing chemotherapeutic treatment to pathological tissue and avoiding surgery related brain tissue damage. Additionally, TMS transiently increases blood-brain barrier permeability, theoretically allowing increased uptake of chemotherapeutic drugs in the target area. This addresses a significant challenge in the treatment of brain cancer, as most cytotoxic drugs have fairly limited ability to pass the blood brain barrier.

The intention of this research project is to investigate the therapeutic potential of focused TMS as an alternative non-invasive source of current induction and thereby means to treat several types of brain cancer with electrochemotherapy.

ELIGIBILITY:
Inclusion Criteria:

* Newly diagnosed and histologically confirmed glioblastoma multiform
* MGMT gene methylation
* If age < 70, eligibility to comply with the Stupp radio chemotherapy regimen
* If age > 70, eligibility for stand alone chemotherapeutic treatment
* Ability to comply with the proposed TMS treatment
* Use of validated anti-conception for fertile female participants in concordance with guidelines provided by the Danish Health and Medicines Authority

Exclusion Criteria:

* Pregnancy or nursing
* Other conditions that may contraindicate the use of transcranial magnetic stimulation
* Implanted pacemaker or metal contraindicating MRI-scan

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 0 (Actual)
Dates: Start 2015-01; Primary Completion 2018-01 (Estimated); Study Completion 2019-05-31 (Actual)

PRIMARY OUTCOMES:
Time to death | 3 years
  Time from onset primary diagnosis until death

SECONDARY OUTCOMES:
Time to progression | 3 years
  Time from diagnosis until radiological tumor progression
Quality of Life | 3 years

CONTACTS AND LOCATIONS:
Overall Officials: Anders R Korshøj, MD, Principal Investigator — Aarhus University Hospital, Department of Neurosurgery